CLINICAL TRIAL: NCT00174395
Title: A Multi-Center, Open-Label, Randomized, Parallel-Group Study of the Effects of Eletriptan 40mg on Mild vs Moderate to Severe Pain Intensity of Migraine in Early Intervention.
Brief Title: A Trial to Study of the Effects of Eletriptan 40mg on Mild vs Moderate to Severe Pain Intensity of Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A1601107
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — eletriptan

INTERVENTIONS:
Drug: eletriptan

SUMMARY:
To evaluate the efficacy of early intervention (dosing within 2 hours of onset of the migraine attack) with eletriptan 40mg on mild versus moderate to severe pain intensity of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine with or without aura according to the recent IHS criteria.
* Migraine headaches must have been present for more than one year.
* History in the last 3 months of 1 to 4 acute attacks of migraine headache per month.

Exclusion Criteria:

* Subjects with current or past history of coronary artery disease.
* Pregnant or breastfeeding women.
* Subjects who have chronic daily headaches.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2005-03; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To evaluate pain free response at 2 hours with eletriptan 40mg in mild pain compared to moderate to severe pain intensity of migraine in early intervention.

SECONDARY OUTCOMES:
To demonstrate the efficacy of early intervention with eletriptan 40mg on mild compared to moderate to severe migraine pain include the following clinical outcomes: pain-free at 0.5, 1, 1.5, 4 and 24 hours; sustained pain-free, migraine recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- Canada (33):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Chilliwack, British Columbia
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, Langley, British Columbia
  - Pfizer Investigational Site, North Vancouver, British Columbia
  - Pfizer Investigational Site, Penticton, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Bathurst, New Brunswick
  - Pfizer Investigational Site, Moncton, New Brunswick
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Truro, Nova Scotia
  - Pfizer Investigational Site, Bolton, Ontario
  - Pfizer Investigational Site, Brampton, Ontario
  - Pfizer Investigational Site, Corunna, Ontario
  - Pfizer Investigational Site, Fort Erie, Ontario
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Markham, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, Niagara Falls, Ontario
  - Pfizer Investigational Site, Woodstock, Ontario
  - Pfizer Investigational Site, Montague, Prince Edward Island
  - Pfizer Investigational Site, Cowansville, Quebec
  - Pfizer Investigational Site, Drummondville, Quebec
  - Pfizer Investigational Site, Granby, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Sainte-Julie, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Regina, Saskatchewan
  - Pfizer Investigational Site, Mount Pearl

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1601107&StudyName=A+Trial+to+Study+of+the+Effects+of+Eletriptan+40mg+on+Mild+vs+Moderate+to+Severe+Pain+Intensity+of+Migraine